CLINICAL TRIAL: NCT02598843
Title: Functional Outcomes After Conservative Management of the Acutely Ruptured Achilles Tendon in the Under 60 Age Group. A Randomised Controlled Trial Comparing Standard Conservative Management With Accelerated Rehabilitation Using a Moon Boot
Brief Title: Standard Non Operative Treatment Versus Accelerated Rehabilitation of Achilles Tendon Ruptures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Lothian (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRAS ID 89061
Record Dates: First submitted 2015-10-15; First posted 2015-11-06 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Rupture of Achilles Tendon

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard treatment protocol (Active Comparator): Cast immobilisation with 4 weeks in equinus cast (non-weight bearing) followed by 4 weeks in semi-equinus cast (non-weightbearing) and 2 weeks in neutral cast (full weightbearing). At this point, the cast is removed and patients mobilise fully weightbearing for a further 2 weeks out of cast, with internal shoe insert heel raise. Commence physiotherapy at 10 weeks, when cast removed.
  Interventions: Other: Standard treatment protocol
- Accelerated rehabilitation (Experimental): 4 weeks in Ossur rebound walking boot with 2 heel wedges (3cm), 2 weeks in Ossur rebound walking boot with 1 heel wedge (1.5cm) and 2 weeks in Ossur rebound walking boot with no heel wedges (neutral position). Fully weightbearing throughout. Commence physiotherapy at 8 weeks.
  Interventions: Other: Accelerated Rehabilitation

INTERVENTIONS:
Other: Standard treatment protocol — Cast Protocol 4 weeks in Full Equinus cast - Non Weight Bearing (NWB) with axillary crutches; 4 weeks in Semi-Equinus cast NWB with axillary crutches; 2 weeks in neutral cast - Full Weight Bearing (FWB); 2 weeks FWB out of cast, with shoe insert heel raise.
  Followed by course of physiotherapy
  Arms: Standard treatment protocol
Other: Accelerated Rehabilitation — 4 weeks in Ossur Rebound walking boot with 3cm heel raise, worn continuously including in bed. Weight bearing as tolerated (WBAT)/FWB - crutches for balance; 2 weeks in Rebound walking boot with 1.5cm heel raise (WBAT/FWB - crutches for balance; 2 weeks in Rebound walking boot with foot in neutral. At 8 weeks, remove boot and allow FWB out of boot.
  At 8 weeks after initiation of treatment, physiotherapy is commenced.
  Arms: Accelerated rehabilitation

SUMMARY:
The purpose of this study is to directly compare traditional plaster treatment with early weightbearing in a walking boot for the non operative treatment of acute achilles tendon rupture.

DETAILED DESCRIPTION:
This injury has traditionally been treated in a plaster cast applied to the leg for a period of 10 weeks which allows the tendon to heal, or by an operation to repair the tendon. Research undertaken in the investigators department has shown that patients treated with surgery or with a plaster had similar chance of re-rupture of the tendon after treatment and gain a similar recovery. The investigators therefore now manage these injuries in a plaster.

More recently, further research has shown that a new type of non-surgical rehabilitation programme, which is quicker than the traditional non-surgical programme, gave a tendon re-rupture rate that was similar to that after surgical treatment. This new rehabilitation programme uses a walking boot fitted with a heel-raise (instead of the traditional plaster). The potential benefit of this quicker rehabilitation programme is that it allows the patient to put weight through the leg immediately, whereas patients treated with the traditional plaster cast non-surgical treatment cannot weight bear (this means that they are kept non-weightbearing and therefore have to use crutches) for the first 8 weeks. The time spent in the walking boot in this new, quicker rehabilitation programme is 8 weeks while that spent in plaster is 10 weeks. This new non-surgical, quicker rehabilitation programme is referred to as the accelerated non-surgical programme hereafter. There are no known increased risks with the accelerated rehabilitation programme.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 16-60 years old with an acute rupture of the Achilles tendon

Exclusion Criteria:

* Patients who do not have an acute rupture (ie. delayed presentation >2 weeks)
* Patients who present with a re-rupture of a previously treated Achilles tendon
* Patients from outside the Lothian (local treatment) area who are unwilling to attend follow-up at the study institution.
* Latex allergy.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 140 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2019-07-03 (Actual); Study Completion 2019-07-03 (Actual)

PRIMARY OUTCOMES:
SMFA (Short Musculoskeletal Function Assessment Questionnaire) | final followup/one year
  46 question score. Patients are asked to tick boxes labelled between 1 (indicating good function/no problems) and 5 (poor function/significant problems) for each question and the responses are used to calculate a "dysfunction index", a "bother index" and an "overall SMFA score". These will be reported for each group with measure of central tendency (mean/median) and standard deviations/interquartile range.

SECONDARY OUTCOMES:
SMFA (Short Musculoskeletal Function Assessment Questionnaire) | At the initial review, upon enrolment in the study, patients are asked to complete the questionnaire detailing their immediate pre-injury status (ie status one day before injury). Then reassessed at 26 weeks.
  46 question score. Patients are asked to tick boxes labelled between 1 (indicating good function/no problems) and 5 (poor function/significant problems) for each question and the responses are used to calculate a "dysfunction index", a "bother index" and an "overall SMFA score". These will be reported for each group with measure of central tendency (mean/median) and standard deviations/interquartile range.
Incidence of thromboembolic events | 1 year
  Incidence of radiologically confirmed thromboembolic events within one year of injury is to be reported for each group.
Ankle and subtalar motion | 10, 26 and 52 weeks
  Ankle motion is to be measured using a goniometer for each patient while subtalar motion is to be clinically assessed. Range of motion will be reported for each group as measure of central tendency (median or mean) and standard deviation or interquartile range.
Calf circumference | 10, 26 and 52 weeks
  Measured in centimetres at a point 11 centimetres below the tibial tuberosity. Both sides are measured and the affected (injured) side is compared to the unaffected (uninjured) side for each patient, yielding a relative calf circumference for the affected side. Relative circumference can then be compared across the two groups and reported for each group as a measure of central tendency along with standard deviation/interquartile range..
Visual Analogue Score (VAS) for pain | Initial review, 4,8,10,26,52 weeks.
  VAS scored between 0 and 10. Patients asked to circle an integer between 0 and 10 to indicate their pain level, with 0 indicating no pain and 10 indicating severe pain. Scores to be reported for each group (arm of trial) as measure of central tendency (mean/median) and standard deviations/interquartile range.
Foot and Ankle Outcomes Questionnaire | At the initial review, upon enrolment in the study, patients are asked to complete the questionnaire detailing their immediate pre-injury status (ie status one day before injury). Then reassessed at 26 and 52 weeks.
  American Academy of Orthopaedic Surgeons (AAOS) questionnaire (August 2005 version based on version 2.0 Foot and Ankles Outcomes Instrument. This consists of 25 questions with patients asked to indicate the answer that best applies to their situation. Responses are used to calculate a score and scores for each group will be reported as a measure of central tendency (median/mean) with standard deviations/interquartile ranges.
Achilles Tendon Total Rupture Score (ATRS) | At the initial review, upon enrolment in the study, patients are asked to complete the questionnaire detailing their immediate pre-injury status (ie status one day before injury). Then reassessed at 26 and 52 weeks
  This is a validated score consisting of 10 questions scored 0 to 10 (whole numbers only) with 0 indicating no limitation and 10 indicating maximal limitation. Data to be analysed and presented as measure of central tendency (median/mean) and standard deviations/interquartile ranges for patients in each group.
Return to work. | 10,26,52 weeks.
  Time to initial return to work activity measured in days from date of injury. To be reported as the measure of central tendency (mean or median) and standard deviation or interquartile range, for each group (arm of trial). Patients will be asked whether they have returned to work when reviewed at each of the review timepoints listed above, until they answer in the affirmative.
Return to driving or public transport. | 10,26,52 weeks.
  Time to initial return to driving (or use of public transport if non-driver), measured in days from date of injury. To be reported as the measure of central tendency (mean or median) and standard deviation or interquartile range, for each group (arm of trial). Patients will be asked whether they have returned to these activities when reviewed at each of the review timepoints listed above, until they answer in the affirmative.
Return to sport. | 10,26,52 weeks.
  Time to initial return to sporting activity (if applicable) measured in days from date of injury. To be reported as the measure of central tendency (mean or median) and standard deviation or interquartile range, for each group (arm of trial). Patients will be asked whether they have returned to sporting activities when reviewed at each of the review timepoints listed above, until they answer in the affirmative.
Achilles tendon rerupture rate | 1 year
  Number of achilles tendon re-ruptures occuring in each group up to one year after injury.
EQ-5D Index and EQ-5D VAS | Pre-injury and post-injury (completed at initial review), 26 weeks and 52 weeks
  The EQ-5D-5L consists of an EQ-5D index, calculated from scores for 5 domains (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) and the index ranges from -1 to +1. The EQ-5D visual analog scale (VAS) asks patients to self-rate their health state on a scale between 0 and 100. Data to be analysed and presented as measure of central tendency (median/mean) and standard deviations/interquartile ranges for patients in each group. This data is collected for the final 41 patients in this study.
Satisfaction Question | 10, 16, 26 and 52 weeks
  Patients asked "How satisfied are you with your treated ankle?". They must choose one of "Very satisfied"/"satisfied"/"neither satisfied nor dissatisfied"/"dissatisfied"/"very dissatisfied". Responses to be analysed as dichotomous data and ordinal data. This data is collected for the final 41 patients in this study.
Patient Preference question | 16 weeks
  Patients asked "Did you have a preference for treatment type for your Achilles tendon injury?" (Choose one of: YES / NO). If Yes, then which modality would you have preferred? (choose one of CAST / BOOT ). Data will be cross tabulated for statistical analysis. This data is collected for the final 41 patients in this study.
Achilles Tendon Total Rupture Score (ATRS) | Post-injury (completed at initial review)
  As above. An additional time point (post-injury), to be completed at the initial review, was added for the final 41 patients in this study.
SMFA (Short Musculoskeletal Function Assessment Questionnaire) | Post-injury (completed at initial review)
  As above. An additional time point (post-injury), to be completed at the initial review, was added for the final 41 patients in this study.
Foot and Ankle Outcomes Questionnaire | Post-injury (completed at initial review)
  As above. An additional time point (post-injury), to be completed at the initial review, was added for the final 41 patients in this study.

CONTACTS AND LOCATIONS:
Overall Officials: Leela Biant, BSc (Hons) MBBS FRSCEd MSres, Principal Investigator — University of Manchester
Locations (1):
- Royal Infirmary Edinburgh, Edinburgh, Lothian, United Kingdom

REFERENCES:
- [Derived] Maempel JF, Clement ND, Duckworth AD, Keenan OJF, White TO, Biant LC. A Randomized Controlled Trial Comparing Traditional Plaster Cast Rehabilitation With Functional Walking Boot Rehabilitation for Acute Achilles Tendon Ruptures. Am J Sports Med. 2020 Sep;48(11):2755-2764. doi: 10.1177/0363546520944905. Epub 2020 Aug 20. PMID 32816521